CLINICAL TRIAL: NCT00278681
Title: An Effectiveness Trial Examining the Addition of Zinc to the Current Case Management Package of Diarrhoea in a Primary Health Care Setting. Phase I
Brief Title: Effectiveness of Adding Zinc to the Current Case Management Package of Diarrhea in a Primary Health Care Setting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Society for Applied Studies (Other)
Collaborators: Johns Hopkins University (Other); World Health Organization (Other)
Responsible Party: Nita Bhandari, Society for Applied Studies, New Delhi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRN-A-96-90006-00; 77955
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-07

CONDITIONS: Diarrhea; Hospitalization
Keywords: zinc; diarrhea; hospitalization; programme
MeSH Terms: conditions — Diarrhea | interventions — Zinc; ORALIT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): Zinc and ORS
  Interventions: Drug: Zinc and ORS

INTERVENTIONS:
Drug: Zinc and ORS — One strip containing 14 dispersible zinc tablets (20 mg each) along with 2 ORS packets were prescribed to all children aged 1 month to 5 years visiting that channel with diarrhea.
  Infants aged less than 6 months were advised half a zinc tablet in a teaspoonful of breast milk; older children were advised 1 tablet in breast milk or clean water.

SUMMARY:
Use of zinc in diarrhea may be an effective intervention to reduce hospitalizations and child mortality as it could reach the most vulnerable children in a community and reduce severity of not only diarrhea but also of associated infections. It might also potentially reduce antibiotic use.

We conducted a pilot study prior to conducting a community based controlled effectiveness trial to assess whether addition of zinc as a therapeutic modality for diarrhea delivered through existing channels, reduces visits to health care providers, antibiotic and other drug use, and increases ORS use during diarrhea.

DETAILED DESCRIPTION:
The pilot study was conducted in a primary health centre (population ~33000) in Faridabad district of the state of Haryana in India. Formative research identified perceptions of caregivers regarding childhood diarrhea, causation and management, care seeking sources and caregivers expectations from healthcare providers. Caregivers in households with children under 5 years old were interviewed in a cross sectional survey to ascertain family characteristics, ORS prescription and use rates, drug prescription rates by healthcare providers and other variables of interest.

In partnership with the local government, channels for distribution of zinc and ORS packets were defined. The channels included physicians (at PHC and private practitioners), auxiliary nurse midwives (ANMs) and Anganwadi workers (AWWs)of the Integrated Child Development Services (ICDS) scheme. Recommendations were developed and translated into local vernacular. A poster, which incorporated the recommendations and pictures of zinc strip and ORS packets, was designed. These posters were put up at different places in the study area. All channels were trained and provided with the supplies of zinc strips and ORS packets except the private practitioners who received only zinc strips and advised caregivers to take ORS packets from government channels. Effectiveness of this pilot program was assessed through 2 cross sectional surveys, 3 and 6 months post training.

The cross sectional surveys revealed that the prescription of syrups, tablets, powders and injections during diarrhea and cost of treatment decreased significantly. Prescription and use of ORS increased markedly. Zinc tablets were prescribed and used in about half the episodes 6 months after start of intervention. It was feasible to train various government and community channels to promote zinc as treatment of acute diarrhea through the primary health care system.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 5 years with diarrhea

Exclusion Criteria:

* Illness requiring hospitalization (referral)

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2364 (Actual)
Dates: Start 2003-08; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
- Reduction in antibiotics and other drugs use during diarrheal illnesses | August 2003 to August 2004
- Increase in ORS use during diarrhea | August 2003 to August 2004
- Reduction in hospitalizations; all cause and diarrhea related | August 2003 to August 2004

CONTACTS AND LOCATIONS:
Overall Officials: Nita Bhandari, PhD, Principal Investigator — Society for Applied Studies
Locations (1):
- Society for Applied Studies, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Result] Bhandari N, Mazumder S, Taneja S, Dube B, Black RE, Fontaine O, Mahalanabis D, Bhan MK. A pilot test of the addition of zinc to the current case management package of diarrhea in a primary health care setting. J Pediatr Gastroenterol Nutr. 2005 Nov;41(5):685-7. doi: 10.1097/01.mpg.0000182799.69675.92. PMID 16254536